CLINICAL TRIAL: NCT05774951
Title: CAMBRIA-1: A Phase III, Open-Label, Randomised Study to Assess the Efficacy and Safety of Extended Therapy With Camizestrant (AZD9833, a Next Generation, Oral Selective Estrogen Receptor Degrader) Versus Standard Endocrine Therapy (Aromatase Inhibitor or Tamoxifen) in Patients With ER+/HER2- Early Breast Cancer and an Intermediate or High Risk of Recurrence Who Have Completed Definitive Locoregional Therapy and at Least 2 Years of Standard Adjuvant Endocrine-Based Therapy Without Disease Recurrence
Brief Title: A Study of Camizestrant in ER+/HER2- Early Breast Cancer After at Least 2 Years of Standard Adjuvant Endocrine Therapy
Acronym: CAMBRIA-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8531C00002; 2022-501024-20-00 (Other: EMA - CTIS)
Record Dates: First submitted 2023-02-16; First posted 2023-03-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer, Early Breast Cancer
Keywords: ER+; HER2-; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833; Tamoxifen; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 1:1 ratio to one of the following arms:
  * Arm A: Continue standard ET of investigator's choice (aromatase inhibitors [AI; exemestane, letrozole, anastrozole] or tamoxifen)
  * Arm B: Camizestrant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: standard endocrine therapy of investigator´s choice (Active Comparator): Continue standard endocrine therapy of investigator's choice (aromatase inhibitors [AI; exemestane, letrozole, anastrozole] or tamoxifen)
  Interventions: Drug: Tamoxifen; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane
- Arm B: camizestrant (Experimental): Camizestrant
  Interventions: Drug: Camizestrant

INTERVENTIONS:
Drug: Camizestrant — Camizestrant. Experimental. Administered orally
  Other Names: AZD9833
  Arms: Arm B: camizestrant
Drug: Tamoxifen — Tamoxifen. Comparator. Administered per local approved label
  Arms: Arm A: standard endocrine therapy of investigator´s choice
Drug: Anastrozole — Anastrozole. Comparator. Administered per local approved label
  Arms: Arm A: standard endocrine therapy of investigator´s choice
Drug: Letrozole — Letrozole. Comparator. Administered per local approved label
  Arms: Arm A: standard endocrine therapy of investigator´s choice
Drug: Exemestane — Exemestane. Comparator. Administered per local approved label
  Arms: Arm A: standard endocrine therapy of investigator´s choice

SUMMARY:
This is a Phase III open-label study to assess if camizestrant improves outcomes compared to standard endocrine therapy in patients with ER+/HER2 - early breast cancer with intermediate or high risk for disease recurrence who completed definitive locoregional therapy (with or without chemotherapy) and standard adjuvant endocrine therapy (ET) for at least 2 years and up to 5 years. The planned duration of treatment in either arm of the study is 60 months.

DETAILED DESCRIPTION:
This is a Phase III open-label study to assess if camizestrant improves outcomes compared to standard endocrine therapy in patients with ER+/HER2 - early breast cancer who completed definitive locoregional therapy (with or without chemotherapy) and standard adjuvant endocrine therapy (ET) for at least 2 years and up to 5 years. The planned duration of treatment in either arm of the study is 60 months. The eligible patients must have intermediate or high risk of recurrence, as defined by specified clinical and biologic criteria. Prior use of CDK4/6 inhibitors is permitted. The primary endpoint of the study is Invasive breast cancer-free survival (IBCFS) and main secondary endpoints include Invasive disease-free survival (IDFS), Distant relapse-free survival (DRFS), Overall survival (OS), Safety and Clinical Outcome Assessments (COAs).

Patients will be followed for 10 years from randomization of the last patient.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men, ≥18 years at the time of screening (or per national guidelines)
* Histologically confirmed ER+/HER2- early-stage resected invasive breast cancer with high or intermediate risk of recurrence, based on clinical-pathological risk features, as defined in the protocol.
* Completed adequate (definitive) locoregional therapy (surgery with or without radiotherapy) for the primary breast tumour(s), with or without (neo)adjuvant chemotherapy
* Completed at least 2 years but no more than 5 years (+3 months) of adjuvant ET (+/- CDK4/6 inhibitor)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Adequate organ and marrow function

Exclusion criteria:

* Inoperable locally advanced or metastatic breast cancer
* Pathological complete response following treatment with neoadjuvant therapy
* History of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix or considered at very low risk of recurrence per investigator judgement) unless in complete remission with no therapy for a minimum of 5 years from the date of randomisation
* Any evidence of severe or uncontrolled systemic diseases which, in the investigator's opinion precludes participation in the study or compliance
* Known LVEF <50% with heart failure NYHA Grade ≥2.
* Mean resting QTcF interval >480 ms at screening
* Concurrent exogenous reproductive hormone therapy or non-topical hormonal therapy for non-cancer-related conditions
* Any concurrent anti-cancer treatment not specified in the protocol with the exception of bisphosphonates (e.g. zoledronic acid) or RANKL inhibitors (eg, denosumab)
* Previous treatment with camizestrant, investigational SERDs/investigational ER targeting agents, or fulvestrant
* Currently pregnant (confirmed with positive serum pregnancy test) or breastfeeding
* Patients with known hypersensitivity to active or inactive excipients of camizestrant or drugs with a similar chemical structure or class to camizestrant. In pre-/peri-menopausal female and male patients, known hypersensitivity or intolerance to LHRH agonists, that would preclude the patient from receiving any LHRH agonist

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4300 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-04-20 (Estimated); Study Completion 2036-05-29 (Estimated)

PRIMARY OUTCOMES:
Invasive breast cancer-free survival (IBCFS) | Up to 10 years
  IBCFS is defined as time from randomisation until date of first occurrence of:
  * Invasive ipsilateral breast tumour recurrence (invasive IBTR)
  * Locoregional invasive breast cancer recurrence
  * Distant recurrence
  * Invasive contralateral breast cancer
  * Death attributable to any cause.

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) | Up to 10 years
  IDFS is defined as time from randomisation until date of first occurrence of one of the following events:
  * Invasive ipsilateral breast tumor recurrence (invasive IBTR)
  * Locoregional invasive breast cancer recurrence
  * Distant recurrence
  * Invasive contralateral breast cancer
  * Second primary non-breast invasive cancer
  * Death attributable to any cause.
Distant relapse-free survival (DRFS) | Up to 10 years
  DRFS is defined as time from randomisation until date of first distant recurrence or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 10 years
  OS is defined as time from randomisation until death from any cause.
Incidence and Severity of Adverse Events, with Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0) | Until 28 days after the final dose of study treatment (up to 5 years)
Absolute and percent change from baseline in Clinical Laboratory Parameters | Until 28 days after the final dose of study treatment (up to 5 years)
Absolute and percent change from baseline in Vital Sign Parameters | Until 28 days after the final dose of study treatment (up to 5 years)
Number of participants with abnormal physical examinations | Until 28 days after the final dose of study treatment (up to 5 years)
Change from baseline of arthralgia as measured by the EORTC-IL-194 (European Organisation for Research and Treatment of Cancer) item 10. EORTC-IL-194 uses 0 - 4 scale (higher score is worse) | Until 28 days after the final dose of study treatment (up to 5 years)
Change from baseline of hot flush as measured by the EORTC-IL-194 item 4. EORTC-IL-194 uses 0 - 4 scale (higher score is worse) | Until 28 days after the final dose of study treatment (up to 5 years)
Change from baseline of vaginal dryness as measured by the EORTC-IL-194 item 15. EORTC-IL-194 uses 0 - 4 scale (higher score is worse) | Until 28 days after the final dose of study treatment (up to 5 years)
Proportion of patients experiencing each level of symptomatic AEs of arthralgia as measured by the EORTC-IL-194 item 10. EORTC-IL-194 uses 0 - 4 scale (higher score is worse) | Until 28 days after the final dose of study treatment (up to 5 years)
Proportion of patients experiencing each level of symptomatic AEs of hot flush as measured by the EORTC-IL-194 item 4. EORTC-IL-194 uses 0 - 4 scale (higher score is worse) | Until 28 days after the final dose of study treatment (up to 5 years)
Proportion of patients experiencing each level of symptomatic AEs of vaginal dryness as measured by the EORTC-IL-194 item 15. EORTC-IL-194 uses 0 - 4 scale (higher score is worse) | Until 28 days after the final dose of study treatment (up to 5 years)
Change from baseline and TTD (time to deterioration ) of health-related QoL (quality of life) as measured by the 2 global QoL items from the EORTC-QLQ-C30 items 11 and 12. EORTC-QLQ-C30 uses 0 - 4 scale (higher score is worse) | Until 28 days after the final dose of study treatment (up to 5 years)
Pharmacokinetics (PK) | Until 6 months from treatment start
  • Plasma concentrations of camizestrant pre-dose (Ctrough)( trough concentration)

CONTACTS AND LOCATIONS:
Locations (555):
- United States (113):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Chandler, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Concord, California
  - Research Site, Corona, California
  - Research Site, Fountain Valley, California
  - Research Site, Greenbrae, California
  - Research Site, Los Alamitos, California
  - Research Site, Palo Alto, California
  - Research Site, San Diego, California
  - Research Site, Whittier, California
  - Research Site, Aurora, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Plantation, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Brewer, Maine
  - Research Site, Scarborough, Maine
  - Research Site, Frederick, Maryland
  - Research Site, Glenn Dale, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Hyannis, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Independence, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Laconia, New Hampshire
  - Research Site, Belleville, New Jersey
  - Research Site, Farmington, New Mexico
  - Research Site, Santa Fe, New Mexico
  - Research Site, East Syracuse, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Clairton, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, State College, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Lancaster, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Aberdeen, South Dakota
  - Research Site, Mitchell, South Dakota
  - Research Site, Pierre, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Yankton, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Denton, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Reston, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Appleton, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Ciudad Autónoma Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Salta
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
  - Research Site, Viedma
- Australia (8):
  - Research Site, Birtinya
  - Research Site, Brighton
  - Research Site, Concord
  - Research Site, Nedlands
  - Research Site, Randwick
  - Research Site, Tweed Heads
  - Research Site, Waratah
  - Research Site, Wendouree
- Austria (12):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Kufstein
  - Research Site, Linz
  - Research Site, Ried
  - Research Site, Sankt Veit an der Glan
  - Research Site, Steyr
  - Research Site, Vienna
  - Research Site, Vöcklabruck
  - Research Site, Wein
  - Research Site, Wels
- Belgium (10):
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mons
  - Research Site, Ottignies
  - Research Site, Wilrijk
  - Research Site, Yvoir
- Brazil (23):
  - Research Site, Alfenas
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Chapecó
  - Research Site, Cuiabá
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Lajeado
  - Research Site, Londrina
  - Research Site, Natal
  - Research Site, Niterói
  - Research Site, Piracicaba
  - Research Site, Porto Alegre
  - Research Site, Pouso Alegre
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Taubaté
  - Research Site, Três Lagoas
  - Research Site, Vitória
- Bulgaria (4):
  - Research Site, Dobrich
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Vratsa
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Barrie, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
- Chile (7):
  - Research Site, Concepción
  - Research Site, La Serena
  - Research Site, Port Montt
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (43):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Dalian
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huangpu District
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Liuchow
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Neijiang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shaoguan
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suining
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wuhan
  - Research Site, Xiangfan
  - Research Site, Xining
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Yanji
  - Research Site, Yantai
  - Research Site, Zhengzhou
- Colombia (8):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Floridablanca
  - Research Site, Medellín
  - Research Site, Montería
  - Research Site, Pereira
  - Research Site, Valledupar
- Czechia (5):
  - Research Site, Hořovice
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Pragues
  - Research Site, Příbram
- France (31):
  - Research Site, Angers
  - Research Site, Argenteuil
  - Research Site, Avignon
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Caen
  - Research Site, Cholet
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Epagny Metz-Tessy
  - Research Site, Lille
  - Research Site, Lorient
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Plerin SUR MER
  - Research Site, Poitiers
  - Research Site, Quimper
  - Research Site, Rennes
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Suresnes
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Villejuif
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (31):
  - Research Site, Aachen
  - Research Site, Augsburg
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Deggendorf
  - Research Site, Dessau
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Eggenfelden
  - Research Site, Esslingen am Neckar
  - Research Site, Georgsmarienhütte
  - Research Site, Gütersloh
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Landshut
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Memmingen
  - Research Site, München
  - Research Site, Ravensburg
  - Research Site, Rüsselsheim am Main
  - Research Site, Stralsund
  - Research Site, Torgau
  - Research Site, Trier
  - Research Site, Ulm
  - Research Site, Velbert
  - Research Site, Wiesbaden
  - Research Site, Worms
  - Research Site, Wuppertal
- Greece (6):
  - Research Site, Athens
  - Research Site, Chaïdári
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Rio
  - Research Site, Thessaloniki
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szekszárd
  - Research Site, Szolnok
- India (15):
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Bhubaneswar
  - Research Site, Hubli
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Thane
  - Research Site, Visakhapatnam
  - Research Site, West Bengal
- Israel (9):
  - Research Site, Afula
  - Research Site, Ashdod
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (14):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Grosseto
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Turin
- Japan (30):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Ōita
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Malaysia (7):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Malacca
  - Research Site, Sabak Bernam
- Mexico (10):
  - Research Site, Aguascalientes
  - Research Site, Alc. Cuauhtémoc
  - Research Site, Colonia Lindavista
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, San Luis Potosí City
  - Research Site, Toluca
  - Research Site, Veracruz
- Netherlands (5):
  - Research Site, Dirksland
  - Research Site, Geleen
  - Research Site, Groningen
  - Research Site, Hoofddorp
  - Research Site, Rotterdam
- Peru (5):
  - Research Site, Arequipa
  - Research Site, Callao
  - Research Site, La Libertad
  - Research Site, Lima
  - Research Site, Trujillo
- Philippines (5):
  - Research Site, Bacolod
  - Research Site, Cebu
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Grudziądz
  - Research Site, Koszalin
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Poznan
  - Research Site, Racibórz
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wieliszew
- Portugal (7):
  - Research Site, Amadora
  - Research Site, Braga
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Romania (11):
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Floreşti
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Sibiu
  - Research Site, Timișoara
- Serbia (6):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Valjevo
  - Research Site, Zrenjanin
- Research Site, Singapore, Singapore
- South Africa (7):
  - Research Site, Bloemfontein
  - Research Site, eManzimtoti
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Pietermaritzburg
  - Research Site, Pretoria
  - Research Site, Soweto
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Donggu
  - Research Site, Goyang-si
  - Research Site, Jeonnam
  - Research Site, Seongbuk-Gu
  - Research Site, Seoul
- Spain (34):
  - Research Site, A Coruña
  - Research Site, Albacete
  - Research Site, Alcoy
  - Research Site, Alicante
  - Research Site, Alzira
  - Research Site, Badajoz
  - Research Site, Badalona
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Cáceres
  - Research Site, Elche(Alicante)
  - Research Site, Galdakao
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Jerez de La Frontera (Cádiz)
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Leganés
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Manresa
  - Research Site, Murcia
  - Research Site, Oviedo
  - Research Site, Parla
  - Research Site, Port de Sagunt
  - Research Site, Reus
  - Research Site, Salamanca
  - Research Site, San Sebastián
  - Research Site, Sant Joan d'Alacant
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Teruel
  - Research Site, Toledo
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Phisanulok
  - Research Site, Phitsanulok
  - Research Site, Rachathewi
  - Research Site, Songkhla
- Turkey (Türkiye) (7):
  - Research Site, Ankara
  - Research Site, Aydin
  - Research Site, Bursa
  - Research Site, Dinar
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Samsun
- United Kingdom (14):
  - Research Site, Brighton
  - Research Site, Burton-on-Trent
  - Research Site, Cambridge
  - Research Site, Derby
  - Research Site, Edinburgh
  - Research Site, Guildford
  - Research Site, Ipswich
  - Research Site, Keighley
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Peterborough
  - Research Site, Stoke-on-Trent
  - Research Site, Sutton
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Hamilton EP, Loibl S, Bachelot T, Gnant M, Niikura N, Park YH, Tolaney SM, Pistilli B, Rastogi P, Saini KS, Gioni I, Johnston S, Nunes R, Quintana A, Stuart M, Syta E, Walding A, Klinowska T, Mayer IA. CAMBRIA-1 & CAMBRIA-2 phase III trials: camizestrant versus standard endocrine therapy in ER+/HER2- early breast cancer. Future Oncol. 2025 Mar;21(7):795-806. doi: 10.1080/14796694.2025.2459548. Epub 2025 Feb 27. PMID 40017004
- See also: Description: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/394222